CLINICAL TRIAL: NCT00605657
Title: Pilot (Phase I-II) Study of Valproic Acid (Depakote) for the Treatment of the Autoimmune Lymphoproliferative Syndrome (ALPS)
Brief Title: Valproic Acid (Depakote[Registered Trademark]) to Treat Autoimmune Lymphoproliferative Syndrome (ALPS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Koneti Rao (NIH)
Responsible Party: Sponsor-Investigator, Koneti Rao, Staff physician, National Institute of Allergy and Infectious Diseases (NIAID)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080053; 08-I-0053 (Other Grant/Funding Number: DIR NIAID)
Record Dates: First submitted 2008-01-15; First posted 2008-01-31 (Estimated); Results first posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-02

CONDITIONS: ALPS; Hypersplenism; Lymphadenopathy
Keywords: ALPS; Valproic Acid; Lymphadenopathy; Splenomegaly; Histone Deacytelase (HDAC) Inhibitor; Autoimmune Lymphoproliferative Syndrome
MeSH Terms: conditions — Hypersplenism; Lymphadenopathy; Splenomegaly; Autoimmune Lymphoproliferative Syndrome | interventions — Valproic Acid; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Valproic acid (Experimental): Single arm study involving oral administration of valproic acid and monitoring of its efficacy by CT scans done before and after the intervention. Blood samples were also obtained to monitor safety labs and biomarkers.
  Interventions: Drug: Valproic Acid; Procedure: CT Scan; Procedure: Blood Sample

INTERVENTIONS:
Drug: Valproic Acid — Oral administration of valproic acid
  Other Names: Depakote
Procedure: CT Scan — CT scans were done before and after treating the patient with valproic acid
  Other Names: Computerized Tomography
Procedure: Blood Sample — Blood samples were collected before and after the intervention to monitor blood counts and biomarkers of ALPS

SUMMARY:
This study will test whether valproic acid (Depakote[Registered Trademark]) can shrink enlarged lymph glands and spleen in patients with autoimmune lymphoproliferative syndrome (ALPS). Depakote has been used for more than 30 years for treating various medical disorders in adults and children, including migraine headaches, seizures and psychiatric disorders. In animal studies, it was effective in shrinking both lymph nodes and spleen in animals with conditions similar to ALPS.

People with ALPS who are between 2 and 70 years of age and who have had an enlarged spleen or lymph glands for at least 1 year may be eligible for this study.

Participants take Depakote as a tablet or liquid or sprinkled on food twice a day for 16 weeks. The drug dose is increased slowly over the first 3 to 4 weeks until the maximum tolerated dose is reached. Blood tests are done at 2, 4, 6, 8 and 10 weeks after starting the drug and 1 week after the drug is stopped to check for treatment side effects. Valproic acid blood levels will be checked during drug escalation, half way through therapy, and just before the end of treatment. A physical examination and CT scan (or ultrasound of the abdomen for patients who cannot undergo CT) are done before starting treatment and at the end of the 16-week treatment period to evaluate the response to treatment.

Patients who tolerate the treatment well and show shrinkage of the lymph glands or spleen may be offered extended treatment for up to 1 year in consultation with their primary physician. During the extended treatment period, blood tests are done at home every 6 to 8 weeks to monitor for drug side effects. Follow up evaluation visits are scheduled at the NIH Clinical Center every 3 months during the extended treatment period and 3, 6, and 12 months after treatment has ended.

DETAILED DESCRIPTION:
The Autoimmune Lymphoproliferative Syndrome (ALPS) is an inherited disease associated with a defect of lymphocyte apoptosis that leads to lymphoproliferation and autoimmunity. Although, there are immunosuppressive treatments for many of its complications, there currently is no safe and effective therapy for this syndrome itself.

Valproic acid has been recently used as a histone deacetylase (HDAC) inhibitor for inducing apoptosis in malignancies and is being incorporated as part of hematology/oncology clinical trials. A pilot study will be conducted on the safety and efficacy of the drug valproic acid (Depakote [R]) for the treatment of ALPS. Twelve subjects with ALPS, will be treated initially for 4 months with twice-daily administration of valproic acid at escalating doses adjusted by weight, with close monitoring of toxicity and side effects including laboratory parameters related to the drug. The effects of valproic acid treatment on lymph node and/or spleen size will be assessed by computerized tomography scan, ultrasound and physical examination. If valproic acid is effective in reducing the size of lymph nodes and/or spleen size as defined in the study design, subjects may be offered the option to continue further therapy with valproic acid for up to 1 year. The effect of treatment on other laboratory features specific to ALPS will also be assessed. Evaluating the effects of valproic acid on these clinical and laboratory parameters will help to determine if this drug demonstrates sufficient activity to warrant study in a larger randomized controlled trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. All subjects must fulfill the published criteria for the diagnosis of ALPS (documented nonmalignant lymphadenopathy and/or splenomegaly of at least 1-year duration; greater than1% TCR alpha/beta+ CD4-CD8- T cells in the peripheral blood). This must include clinically documented lymphadenopathy involving more than 2 nodes in more than 1 regional group of nodes measuring greater than 2cm in size and/or a palpable spleen.
  2. Age greater than or equal to 2 years through less than or equal to 70 years.
  3. Must have a personal primary care physician who is willing to follow the protocol required evaluations during the study period.
  4. Must be willing to sign a consent form.
  5. Patients on immunosuppression (e.g., corticosteroid, mycophenolate mofetil, azathioprine, cyclophosphamide) are eligible if the dose of the immunosuppressive drug has been stable for at least 3 months prior to enrollment and their hematologic parameters do not meet the exclusion criteria (1) as outlined below.

EXCLUSION CRITERIA:

1. A hemoglobin concentration of less than 8 gm/dL, a platelet count of less than 75 K/mm(3), or an absolute neutrophil count of less than 500/mm(3), at study entry.
2. Liver disease determined by an alanine aminotransferase (ALT), aspartate aminotransferase (AST), or bilirubin 2.5 times greater than the upper limit of normal.
3. History of pancreatitis by clinical features and/or laboratory abnormalities in the last 12 months.
4. Renal dysfunction determined by a calculated urine creatinine clearance of less than 70 mL/min/1.73 m(2) in children and less than 60 mL/min in adults, or using the Schwartz formula or Levy formula based on serum creatinine.
5. Patients clinically suspected of suffering from urea cycle disorders will be excluded.
6. Patients with history of seizure disorders and/or those already receiving valproic acid will be excluded.
7. Sensitive to or have ever had an allergic reaction to Depakote.
8. Not able to abstain from alcohol during the length of the study.
9. Pregnancy. Female adults and adolescents who have attained menarche must have a negative pregnancy test at study entry and commit to using an acceptable method of barrier or hormonal contraception (e.g., condoms, diaphragms, oral contraceptives, or long acting progestin agents) if sexually active during the study and for 3 months after the last dose of valproic acid.
10. Lactating mothers who are breast feeding their babies will not be eligible.
11. ALPS patients who have been treated with bone marrow toxic chemotherapy regimens for Non-Hodgkin's lymphoma or other malignancies are not eligible for this pilot study.
12. Unwilling or unable to comply with the need to have periodic blood tests to monitor possible side effects of treatment, or other major requirements of this study will be an exclusion criteria.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koneti Rao, MD, Principal Investigator — DIR, NIAID, NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sneller MC, Straus SE, Jaffe ES, Jaffe JS, Fleisher TA, Stetler-Stevenson M, Strober W. A novel lymphoproliferative/autoimmune syndrome resembling murine lpr/gld disease. J Clin Invest. 1992 Aug;90(2):334-41. doi: 10.1172/JCI115867. PMID 1386609
- [Background] Rao VK, Straus SE. Causes and consequences of the autoimmune lymphoproliferative syndrome. Hematology. 2006 Feb;11(1):15-23. doi: 10.1080/10245330500329094. PMID 16522544
- [Background] Rao VK, Carrasquillo JA, Dale JK, Bacharach SL, Whatley M, Dugan F, Tretler J, Fleisher T, Puck JM, Wilson W, Jaffe ES, Avila N, Chen CC, Straus SE. Fluorodeoxyglucose positron emission tomography (FDG-PET) for monitoring lymphadenopathy in the autoimmune lymphoproliferative syndrome (ALPS). Am J Hematol. 2006 Feb;81(2):81-5. doi: 10.1002/ajh.20523. PMID 16432855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were started on valproic acid at the NIH Clinical Center then followed locally
Groups:
- Valproic Acid: valproic acid administered starting at 10 mg/kg/day in divided doses twice daily x 3 days, increase to 15mg/kg/day x 3 days, increase to 20 mg/kg/day on day 7, increase to 30 mg/kg/day on day 14, maximum dose of 40mg/kg/day on day 21, if tolerated, to achieve plasma level 50-100 mcg/mL.
Period: Overall Study
Arm/Group | Valproic Acid
Started | 5
Completed | 3
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Valproic Acid
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Reduction of lymph node and/or spleen size measured by CT imaging, or physical exam and abdominal ultrasound. A clinical response is defined as a greater than 40% reduction in lymph node size and/or greater than 40% reduction in spleen size. A CT scan with contrast measured lymph node size as well as spleen size.
Time Frame: 3 monthly (12 week) intervals
Measure: Number; unit: participants
Arm/Group | Valproic Acid
Number analyzed (Participants) | 3
participants | 0

2. Secondary Outcome: To Determine Whether the Treatment Alters, in Favorable Directions, Laboratory Markers of ALPS (e.g., Number of DNT Cells, Immunoglobin Levels, Vitamin B12 Levels, IL-10 Levels, Autoantibody Titers, Fas Mediated Apoptosis)
Time Frame: 3 monthly (12 week) intervals
Population: outcome measure not assessed because 0 participants had a response
Arm/Group | Valproic Acid
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Valproic Acid
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproic Acid (N=5)
pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) — not treatment related
low serum IgG (Blood and lymphatic system disorders) | 1 (1) — possibly related to treatment
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproic Acid (N=5)
fever (General disorders) | 2 (2) — unrelated
decreased platelets (Blood and lymphatic system disorders) | 3 (3) — Only probably related in one patient. Other patients had baseline low platelets.
decreased hemoglobin (Blood and lymphatic system disorders) | 3 (3) — unlikely or unrelated in all patients
decreased neutrophil count (Blood and lymphatic system disorders) | 4 (4) — unlikely or unrelated in all cases
hyperglycemia (General disorders) | 1 (1) — unrelated
vomiting (Gastrointestinal disorders) | 1 (1) — vomiting unrelated, due to the flu in one case. Possibly related in other
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — unrelated
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — unrelated
fatigue (General disorders) | 5 (5) — not related in two cases, possibly related in one case.
rhinorrhea (General disorders) | 1 (1) — unrelated
elevated AST (Gastrointestinal disorders) | 2 (2) — one probably related and one unlikely related
elevated ALT (Gastrointestinal disorders) | 1 (1) — probably related
diarrhea (Gastrointestinal disorders) | 1 (1) — possibly related
gastroenteritis (Gastrointestinal disorders) | 1 (1) — possibly related
pruritis (Skin and subcutaneous tissue disorders) | 1 (1) — probably related
leukopenia (Blood and lymphatic system disorders) | 2 (2) — unlikely or unrelated
abdominal pain (Gastrointestinal disorders) | 1 (1) — possibly related
nausea (Gastrointestinal disorders) | 1 (1) — possibly related
elevated alkaline phosphatase (Blood and lymphatic system disorders) | 1 (1) — unrelated
rash (Skin and subcutaneous tissue disorders) | 2 (2) — probably related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes